CLINICAL TRIAL: NCT01348516
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Single/Multiple Dosing, Dose-escalation Clinical Trial to Investigate the Safety, Tolerability, and Pharmacokinetic Characteristics of KM-023 After Oral Administration in Healthy Subjects
Brief Title: Single Ascending Dose (SAD)/Multiple Ascending Dose(MAD) Safety/Pharmacokinetic (PK) Study of KM-023
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kainos Medicine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMCP-023-101
Record Dates: First submitted 2011-05-02; First posted 2011-05-05 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — 3-(3-ethyl-5-isopropyl-2,6-dioxo-1,2,3,6-tetrahydropyrimidine-4-carbonyl)-5-methylbenzonitrile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- KM-023 (Experimental)
  Interventions: Drug: KM-023
- Placebo for KM-023 (Placebo Comparator)
  Interventions: Drug: Placebo for KM-023

INTERVENTIONS:
Drug: KM-023 — -KM-023 is dosed orally via 75 mg tablets. Study doses are 75 mg, 150 mg, 300 mg, and 600 mg QD for 1 (SAD) or 7 (MAD) days.
  Arms: KM-023
Drug: Placebo for KM-023 — -Placebo for KM-023 is dosed orally via Placebo for KM-023 tablets. Study doses are 1, 2, 3, and 4 placebo tablets QD for 1 (SAD) or 7 (MAD) days.
  Arms: Placebo for KM-023

SUMMARY:
The purpose of this study is to investigate the safety and pharmacokinetics of KM-023 after single/multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

* Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB) - approved informed consent prior to performing any of the screening procedures
* Male or female between 20 and 45 years of age at the time of screening, inclusive
* A subject with body weight ≥ 45 kg and body mass index (BMI) between 18.5 and 25 (inclusive). - BMI (kg/m2) = weight (kg) / {height (m)}2
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

1. A subject with a history of allergies to drugs (aspirin, antibiotics, etc.), or history of clinically significant allergies
2. A subject with clinical evidence or history of hepatic (including carrier of hepatitis virus), renal, respiratory, endocrine, neurologic, immunologic, hematologic, oncologic, psychiatric, or cardiovascular disease
3. A subject with a history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug
4. A female subject who is pregnant, nursing mother, or sexually active females (childbearing potential)
5. Patients who are taking any of the following medications; Bepridil, cisapride, midazolam, pimozide, triazolam, Ergot medications (e.g. Wigraine, cafergot, St. John's wort), Phenobarbitol
6. Patients who have previously demonstrated hypersensitivity to Efavirenz or to one of the components of Stocrin or Sustiva
7. A positive Hepatitis B surface antigen or positive Hepatitis C antibody at screening.
8. A positive test for HIV antibody (as per local practice)
9. A subject who has taken any prescribed medication or herbal compounds within 14 days prior to the study drug administration. In addition, a subject who has taken any over-the-counter drug or vitamin supplements within 7 days prior to the study drug administration.
10. A subject who has participated in any other clinical trial either for investigational or marketed drugs within 8 weeks before the study drug administration
11. A subject who has donated or had loss of ≥ 400 mL of blood within 8 weeks prior to start of administration of study drug
12. The value of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) is greater than 1.25 times the upper limit of the reference range.
13. A subject who is unable to abstain from drinking alcoholic beverages throughout the study period.
14. A subject with a history of drug abuse, or a positive urine drug screening test
15. A subject who heavily takes caffeine or caffeine-containing products, or takes grapefruit, grapefruit juice, or grapefruit-containing products
16. A subject who is unable to eat a standardized meal offered by the study center
17. A subject who will be previously assigned to treatment during this study (except those who did not take any study medications)
18. Systolic blood pressure outside the range of 80 to 140 mm Hg, or diastolic blood pressure outside the range of 60 to 85 mm Hg, or heart rate outside the range of 50 to 100 beats per minute (bpm) for females; outside and the range of 45 to 100 beats per minute (bpm) for male subjects. Blood pressure and heart rate should be taken after 10 minutes of rest.
19. The investigator judges the subject not eligible for the study after reviewing clinical laboratory results or other reasons

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety/ Tolerability Evaluation | participants will be followed for the duration of hospital stay, 8-10 days for SAD and 14-16 days for MAD
  -number of subjects with Adverse events, Physical examinations, Vital signs, electrocardiogram (ECG), Laboratory tests (including hematology, chemistry, coagulation, urinalysis), circulating immune complexes (CIC)

SECONDARY OUTCOMES:
Pharmacokinetic Evaluation of KM-023, Area under the plasma concentration versus time curve (AUC) of KM-023 | participants will be followed for the duration of hospital stay, 8-10 days for SAD and 14-16 days for MAD
  -Serial blood samples and urine collections for pharmacokinetic evaluations will be conducted pre-dose through post dose in order to evaluate AUC of KM-023
Pharmacokinetic Evaluation of KM-023, Peak Plasma Concentration (Cmax) of KM-023 | participants will be followed for the duration of hospital stay, 8-10 days for SAD and 14-16 days for MAD
  -Serial blood samples and urine collections for pharmacokinetic evaluations will be conducted pre-dose through post dose in order to evaluate Cmax of KM-023

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Center, Seoul National University Hospital, Seoul, South Korea